CLINICAL TRIAL: NCT04352478
Title: Incidental Cancer in Gallbladder Surgical Specimens Focus on Elderly Patients, Retrospective Analysis of 2389 Patients
Brief Title: Incidental Cancer in Gallbladder Surgical Specimens Focus on Elderly Patients
Status: Completed | Type: Observational
Sponsor: Dr. Ersin Arslan Education and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Uylas, Specialist, Dr. Ersin Arslan Education and Training Hospital
Other Study IDs: 13042020
Record Dates: First submitted 2020-04-13; First posted 2020-04-20 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Pathology
Keywords: cholecystectomy; cholecystitis; cholelithiasis; gallbladder neoplasms; histopathology; surgical procedures
MeSH Terms: conditions — Cholecystitis; Cholelithiasis; Gallbladder Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elder: elderly (≥60 years old).
  Interventions: Diagnostic Test: Histopathological result
- Young: young (<60 years old)
  Interventions: Diagnostic Test: Histopathological result

INTERVENTIONS:
Diagnostic Test: Histopathological result — Incidental gallbladder cancer and other pathology

SUMMARY:
Causes such as long-term stones and polyp are thought to play a role in the etiology of gallbladder cancer. The routine histopathological examination provides the detection of incidental gallbladder cancers. It should be remembered that acute or chronic cholecystitis accompanied by the thicked wall and a prolonged history of gallstones may be the cause of malignancy, especially in elderly patients.

DETAILED DESCRIPTION:
The investigators aimed to incidental gallbladder cancer and compare other pathology results with elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* acute cholecystectomy
* elective cholecystectomy

Exclusion Criteria:

* lack of data
* incidental cholecystectomy,
* cholecystectomy secondary to trauma
* cholecystectomy secondary to malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent cholecystectomy between January 2016 and February 2020 at our hospital
Sampling Method: Non-Probability Sample
Enrollment: 2389 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-13 (Actual)

PRIMARY OUTCOMES:
Rate of Incidental Cancer | 2 or 3 week
  Number of Participants with adenocarcinom

CONTACTS AND LOCATIONS:
Overall Officials: Ufuk Uylas, Principal Investigator — Dr. Ersin Arslan Training and Resource Hospital
Locations (1):
- Dr. Ersin Arslan Training and Resource Hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided